CLINICAL TRIAL: NCT02745522
Title: Can Oxytocin Enhance the Placebo Effect?
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Prof., University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-07
Record Dates: First submitted 2016-03-11; First posted 2016-04-20 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Oxytocin Effect on Memory Performance During Phase 1; Oxytocin Effect on Memory Performance During Phase 2; Oxytocin Effect on Memory Performance During Phase 3; Oxytocin Effect on Memory Performance During Phase 4
Keywords: Placebo effect; Working memory
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Oxytocin (Experimental): Oxytocin nasal spray
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Placebo nasal spray
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin
  Arms: Oxytocin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The current study aimed to investigate whether oxytocin (OXT) had effect on placebo effect.

DETAILED DESCRIPTION:
The current study included three phases to investigate oxytocin effect on placebo effect:

1. In a double-blind, between-subject, placebo controlled design study to investigate the intranasal OXT (24IU) treatment in 66 healthy male subjects using working memory task.
2. In a single-blind(subjects were informed that the treatment was oxytocin), between-subject, placebo controlled design study to investigate the intranasal OXT (24IU) treatment in 53 healthy male subjects using working memory task.They were informed that oxytocin would increase memory perfomance by a female experimenter.
3. In a single-blind(subjects were informed that the treatment was oxytocin), between-subject, placebo controlled design study to investigate the intranasal OXT (24IU) treatment in 53 healthy male subjects using working memory task. But the subjects were told that oxytocin would decrease the performance by the same female experimenter.
4. In a single-blind(subjects were informed that the treatment was oxytocin), between-subject, placebo controlled design study to investigate the intranasal OXT (24IU) treatment in 52 healthy male subjects using working memory task. The subjects were told that oxytocin would increase the performance by a male experimenter.

Memory performance was included as dependant factor. All subjects completed a range of questionnaires measuring personality and affective traits and levels of anxiety: State-Trait Anxiety Inventory (STAI), Beck Depression Inventory (BDI), Interpersonal Trust Scale(ITS).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorder

Exclusion Criteria:

* history of head injury;
* claustrophobia;
* medical or psychiatric illness.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 224 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Memory performance in different phases | 1 hour
  N-back memory performance (accuracy) was included into analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Life Science and Technology, University of Electronic Science and Technology, Chengdu, Sichuan, China